CLINICAL TRIAL: NCT00930904
Title: Attain Ability® Model 4196 Left Ventricular Lead Chronic Performance Post Approval Study
Brief Title: Model 4196 Left Ventricular (LV) Lead Chronic Performance Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 4196 Chronic Performance
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate long-term performance of the 4196 LV Lead. This evaluation is based on the number of lead-related complications occurring during the study compared to the number of leads enrolled in the study. The leads will be followed for 5 years after implant. This study is required by FDA as a condition of approval of the Model 4196 LV Lead and is integrated within the Product Surveillance Registry (PAN Registry).

DETAILED DESCRIPTION:
Model 4196 LV lead complication-free survivability will be summarized.

ELIGIBILITY:
Patients who meet all of the following inclusion criteria and do not meet any of the following exclusion criteria are eligible for enrollment.

Inclusion Criteria

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive an Attain Ability Model 4196 LV lead
* Patient within 30 day post implant enrollment window

Exclusion Criteria

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with a 4196 LV Lead within the past 30 days. All patients must meet Inclusion criteria and none of the Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1847 (Actual)
Dates: Start 2009-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Lead-related complication rate | 5 years

SECONDARY OUTCOMES:
Types of lead-related events | 5 years
Percent of subjects with changes in electrode programming | 5 Years
Percent of fractures with loss of function | 5 years
Mean bipolar pacing threshold | 1 year
Mean pacing threshold and impedance via Tip and Ring unipolar pacing configurations | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: 4196 LV Lead Chronic Performance Study Team, Study Chair — Medtronic
Locations (103):
- United States (91):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Gilbert, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - Downey, California
  - East Palo Alto, California
  - Long Beach, California
  - Salinas, California
  - San Bernardino, California
  - Torrance, California
  - Van Nuys, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Marietta, Georgia
  - Oak Lawn, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Alexandria, Louisiana
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Worcester, Massachusetts
  - Grand Blanc, Michigan
  - Marquette, Michigan
  - Saginaw, Michigan
  - Ypsilanti, Michigan
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Browns Mills, New Jersey
  - Ocean City, New Jersey
  - Parlin, New Jersey
  - West Orange, New Jersey
  - Albuquerque, New Mexico
  - Huntington, New York
  - Utica, New York
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Sayre, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Florence, South Carolina
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Burlington, Vermont
  - Fairfax, Virginia
  - Olympia, Washington
  - Spokane, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Linz, Austria
- Hasselt, Belgium
- Canada (4):
  - Ottawa, Ontario
  - Ste-Foy, Quebec
  - Kingston
  - Toronto
- Marseille, France
- Italy (2):
  - Reggio Emilia
  - Udine
- Netherlands (2):
  - Eindhoven
  - Rotterdam
- Valencia, Spain